CLINICAL TRIAL: NCT07400627
Title: Comparison of the Effectiveness of Ultrasound-Guided Direct and Seldinger Cannulation Techniques in Patients With Anticipated Difficult Radial Artery Cannulation Undergoing Cardiac Surgery
Brief Title: Direct vs. Seldinger Technique for Ultrasound-Guided Difficult Radial Access in Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Professor of Anesthesiology, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AEŞH-EK-2025-221
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Surgery in Adult Patient; Cardiac Surgery; Radial Artery Cannulation; Arterial Cannulation; Radial Artery Catheterization
Keywords: difficult radial artery cannulation; direct technique for radial artery cannulation; Seldinger technique for radial artery cannulation

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Direct Cannulation Technique (Experimental): Patients in this group will undergo radial artery cannulation using the ultrasound-guided direct technique.
  Interventions: Procedure: Ultrasound-Guided Direct Cannulation Technique
- Ultrasound-Guided Seldinger Cannulation Technique (Active Comparator): Patients in this group will undergo radial artery cannulation using the ultrasound-guided Seldinger technique.
  Interventions: Procedure: Ultrasound-Guided Seldinger Cannulation Technique

INTERVENTIONS:
Procedure: Ultrasound-Guided Direct Cannulation Technique — Radial artery cannulation performed using the direct puncture technique (catheter-over-needle) under real-time ultrasound guidance.
  Arms: Ultrasound-Guided Direct Cannulation Technique
Procedure: Ultrasound-Guided Seldinger Cannulation Technique — Radial artery cannulation performed using the Seldinger technique (catheter-over-guide-wire) under real-time ultrasound guidance.
  Arms: Ultrasound-Guided Seldinger Cannulation Technique

SUMMARY:
Radial artery cannulation is a routine procedure for invasive hemodynamic monitoring for patients undergoing cardiovascular surgery patients.

Although ultrasound (USG) guidance is known to improve success rates, there is limited data comparing the efficacy of the 'Direct' versus 'Seldinger' techniques specifically in patients with anticipated difficult radial access.

This study aims to compare the effectiveness of USG-guided Direct cannulation and USG-guided Seldinger techniques in adult patients with anticipated difficult radial arterial cannulation.

DETAILED DESCRIPTION:
Study Protocol and Patient Assessment: Data collection and the procedural intervention will be performed in the preoperative period, prior to the induction of anesthesia. All patients will undergo a modified Allen test. The radial artery site will be selected based on the following hierarchy: preferably the non-dominant hand (unless surgical plan dictates otherwise), an arm with no history of coronary angiography, and the side determined to be easiest for cannulation via ultrasound (USG) assessment.

Ultrasound Assessment and Exclusion: A 12 MHz linear ultrasound probe will be used for all assessments and procedures. Before the intervention, a detailed sonographic evaluation of the radial artery will be recorded, including:

* Artery diameter and wall thickness
* Lumen continuity and flow velocity
* Presence of calcification, vessel irregularity, or tortuosity
* Stenosis (percentage) and plaque characterization (stable/unstable; fibrous/fatty)
* Presence of hematoma, posterior wall injury, or dissection
* Skin- mid radial artery distance Patients with significant stenosis where an appropriate arterial segment matching the cannula diameter and length cannot be identified will be excluded from the study, and cannulation will be performed at an alternative site.

Randomization and Positioning: Patients will be randomized into two groups using a computer-generated random number table:

* Group D (Direct): Cannulation performed using the catheter-over-needle technique.
* Group S (Seldinger): Cannulation performed using the catheter-over-guide-wire technique.

The patient's arm will be abducted, and the wrist will be extended and fixed over a small support. Standard aseptic preparation and draping will be performed.

Procedural Definitions and Outcome Measures: The procedure will be performed under real-time ultrasound guidance. The following time intervals and metrics will be recorded:

* Radial artery cannulation time: Defined as the time elapsed from the initial skin contact of the needle/cannula to the appearance of the radial artery pressure waveform
* Radial artery puncture time: Defined as the time elapsed from the initial skin contact of the needle/cannula to the appearance of blood in the hub Number of puncture: The total number of skin punctures required to achieve successful cannulation.

Number of needle maneuvers: The total number of needle advancements towards the artery

Safety and Follow-up: If arterial cannulation fails, manual compression will be applied to the artery for 5 minutes to prevent hematoma formation. All patients will be monitored for complications (such as hematoma, ischemia, or nerve injury) for 24 hours post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* American Society of Anesthesiologists (ASA) physical status I-IV
* Patients scheduled for cardiovascular surgery requiring invasive arterial monitoring

Exclusion Criteria:

* Patients undergoing emergency surgery
* Coagulation disorders or known coagulopathy
* Presence of an arteriovenous fistula
* Patients in shock or hemodynamically instable
* Patients requiring mechanical circulatory support
* History of Raynaud's phenomenon
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
First-Attempt Cannulation Success Rate | 10 min before anesthesia induction
  The proportion of patients in whom radial artery cannulation is successfully performed (verified by the appearance of the arterial pressure waveform on the monitor) with a single skin puncture

SECONDARY OUTCOMES:
Number of Cannulation Attempts | 10 min before anesthesia induction
  The total number of skin punctures required to achieve successful radial artery cannulation
Radial artery cannulation time | 10 min before anesthesia induction
  Total time elapsed from the initial skin contact with the arterial cannula to the visualization of the arterial waveform on the monitor.
Incidence of Procedure-Related Complications | Postoperative 24th hour
  Evaluation of adverse events associated with the cannulation procedure, including hematoma, arterial dissection, posterior wall injury, nerve injury, or infection

CONTACTS AND LOCATIONS:
Overall Officials: Dilek ÜNAL, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Kader, A. , Kaushal, N. , Shah, R. , Gomulka, M. , Wang, T. and Shulman, S. (2016) A Novel Technique to Maintain Radial Arterial Catheter Position: The Arterial Catheter Stabilizer. Open Journal of Anesthesiology, 6, 193-197. doi: 10.4236/ojanes.2016.612029.
- [Background] Sung JM, Jun YE, Jung YD, Kim KN. Comparison of an Ultrasound-Guided Dynamic Needle Tip Positioning Technique and a Long-Axis In-Plane Technique for Radial Artery Cannulation in Older Patients: A Prospective, Randomized, Controlled Study. J Cardiothorac Vasc Anesth. 2023 Dec;37(12):2475-2481. doi: 10.1053/j.jvca.2023.08.138. Epub 2023 Aug 25. PMID 37741770
- [Background] Mesa BK, Sinha M, Kumar M, Ramchandani S, Dey C, Agrawal N, Khetarpal M. Radial Arterial Cannulation by Ultrasound-Guided Dynamic Needle-Tip Positioning Using the Short-Axis Out-of-Plane Approach Versus the Long-Axis In-Plane Approach: A Randomized Controlled Study. Cureus. 2024 Feb 14;16(2):e54183. doi: 10.7759/cureus.54183. eCollection 2024 Feb. PMID 38496072
- [Background] Nam K, Jeon Y, Yoon S, Kwon SM, Kang P, Cho YJ, Kim TK. Ultrasound-guided radial artery cannulation using dynamic needle tip positioning versus conventional long-axis in-plane techniques in cardiac surgery patients: a randomized, controlled trial. Minerva Anestesiol. 2020 Jan;86(1):30-37. doi: 10.23736/S0375-9393.19.13646-2. Epub 2019 Jun 17. PMID 31213045